CLINICAL TRIAL: NCT01966354
Title: Comparison of Three Techniques for Ultrasound-guided Internal Jugular Cannulation: Long Axis, In-plane Needle v. Short Axis, Out-of-plane Needle v. Oblique Axis, In-plane Needle
Brief Title: Comparison of Three Techniques for Ultrasound-guided Internal Jugular Cannulation
Acronym: OISO-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mikel Batllori (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Mikel Batllori, Mikel Batllori Gaston, MD, Fundacion Miguel Servet
Organization: Fundacion Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI12/00679
Record Dates: First submitted 2013-10-11; First posted 2013-10-21 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-06

CONDITIONS: Ultrasound-guided Internal Jugular Cannulation; Central Venous Access Complications
Keywords: adult; catheterization, central venous; ultrasonography, interventional; evidence-based medicine; cost-benefit analysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Long axis, in-plane needle (Experimental): Ultrasound-guided Internal jugular venous approach
  Long axis, in-plane needle:
  Jugular vein is ultrasonographically visualized in a longitudinal fashion (long axis) and the needle is inserted in the same ultrasound plane, aligned with the longitudinal axis of the transducer.
  Interventions: Procedure: Ultrasound-guided Internal jugular venous approach
- Short axis, out-of-plane needle (Experimental): Ultrasound-guided Internal jugular venous approach
  Short axis, out-of-plane needle:
  Jugular vein is ultrasonographically visualized in a transverse fashion (short axis) and the needle is inserted perpendicular to the longitudinal axis of the transducer (out-of-plane).
  Interventions: Procedure: Ultrasound-guided Internal jugular venous approach
- Oblique axis, in-plane needle (Experimental): Ultrasound-guided Internal jugular venous approach
  Oblique axis, in-plane needle:
  Jugular vein is ultrasonographically visualized in an oblique axis (intermediate view between long and short axis) and the needle is inserted in the same ultrasound plane, aligned with the longitudinal axis of the transducer.
  Interventions: Procedure: Ultrasound-guided Internal jugular venous approach

INTERVENTIONS:
Procedure: Ultrasound-guided Internal jugular venous approach — The physician will use an ultrasound machine to perform an ultrasound-guided internal jugular venous cannulation: the needle and the vein will be visualized in real time in the ultrasound image to make the cannulation process easier and safer.
  In each one of three study arms, however, the ultrasound approach will be different depending on the axis on wich the vein is visualized (longitudinal, transversal or oblique) and the way the needle enters the ultrasound plane (in-plane or out of plane).

SUMMARY:
The purpose of this study is to assess the efficacy and safety of three ultrasound assistance techniques for internal jugular venous cannulation, in terms of cannulation success and prevention of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Indication for internal jugular venous cannulation, previously established by the doctor responsible for the patient´s hospital diagnosis and treatment
* Informed consent for trial participation has been obtained from the patient

Exclusion Criteria:

* Infection signs at or close to puncture site
* Cutaneous erosions or subcutaneous haematoma at or close to puncture site
* History of internal jugular venous cannulation during the past 72 hours (in the same side in which the present cannulation is taking place)
* History of previous surgical interventions on the cannulation site
* Recent cervical trauma with present neck immobilization and without having ruled out eventual cervical spinal injury
* Severe coagulopathy (altered coagulation parameters and active bleeding) which cannot be promptly corrected by platelet, fresh frozen plasma or pharmacologic intervention
* Subcutaneous emphysema with cervical extension
* Agitated or uncooperative patient (including deep sedation)
* Inability to obtain formal informed consent from the patient or his legally authorized representative (in case the patient is legally incompetent to give informed consent)
* Cannulation being performed outside the surgical area or the post-anesthesia care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Batllori, MD, Study Director — Complejo Hospitalario de Navarra, Anesthesiology department
Locations (1):
- Complejo Hospitalario de Navarra, Anesthesiology department, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Eisen LA, Narasimhan M, Berger JS, Mayo PH, Rosen MJ, Schneider RF. Mechanical complications of central venous catheters. J Intensive Care Med. 2006 Jan-Feb;21(1):40-6. doi: 10.1177/0885066605280884. PMID 16698743
- [Background] Maecken T, Grau T. Ultrasound imaging in vascular access. Crit Care Med. 2007 May;35(5 Suppl):S178-85. doi: 10.1097/01.CCM.0000260629.86351.A5. PMID 17446777
- [Background] Karakitsos D, Labropoulos N, De Groot E, Patrianakos AP, Kouraklis G, Poularas J, Samonis G, Tsoutsos DA, Konstadoulakis MM, Karabinis A. Real-time ultrasound-guided catheterisation of the internal jugular vein: a prospective comparison with the landmark technique in critical care patients. Crit Care. 2006;10(6):R162. doi: 10.1186/cc5101. PMID 17112371
- [Background] Milling TJ Jr, Rose J, Briggs WM, Birkhahn R, Gaeta TJ, Bove JJ, Melniker LA. Randomized, controlled clinical trial of point-of-care limited ultrasonography assistance of central venous cannulation: the Third Sonography Outcomes Assessment Program (SOAP-3) Trial. Crit Care Med. 2005 Aug;33(8):1764-9. doi: 10.1097/01.ccm.0000171533.92856.e5. PMID 16096454
- [Background] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984
- [Background] Shojania KG, Duncan BW, McDonald KM, Wachter RM, Markowitz AJ. Making health care safer: a critical analysis of patient safety practices. Evid Rep Technol Assess (Summ). 2001;(43):i-x, 1-668. PMID 11510252
- [Background] Hessel EA 2nd. Con: we should not enforce the use of ultrasound as a standard of care for obtaining central venous access. J Cardiothorac Vasc Anesth. 2009 Oct;23(5):725-8. doi: 10.1053/j.jvca.2009.06.020. No abstract available. PMID 19789059
- [Background] Augoustides JG, Cheung AT. Pro: ultrasound should be the standard of care for central catheter insertion. J Cardiothorac Vasc Anesth. 2009 Oct;23(5):720-4. doi: 10.1053/j.jvca.2009.06.012. Epub 2009 Aug 15. No abstract available. PMID 19686963
- [Background] Blaivas M, Adhikari S. An unseen danger: frequency of posterior vessel wall penetration by needles during attempts to place internal jugular vein central catheters using ultrasound guidance. Crit Care Med. 2009 Aug;37(8):2345-9; quiz 2359. doi: 10.1097/CCM.0b013e3181a067d4. PMID 19531950
- [Background] Moon CH, Blehar D, Shear MA, Uyehara P, Gaspari RJ, Arnold J, Cukor J. Incidence of posterior vessel wall puncture during ultrasound-guided vessel cannulation in a simulated model. Acad Emerg Med. 2010 Oct;17(10):1138-41. doi: 10.1111/j.1553-2712.2010.00869.x. PMID 21069895
- [Background] Stone MB, Moon C, Sutijono D, Blaivas M. Needle tip visualization during ultrasound-guided vascular access: short-axis vs long-axis approach. Am J Emerg Med. 2010 Mar;28(3):343-7. doi: 10.1016/j.ajem.2008.11.022. Epub 2010 Jan 28. PMID 20223394
- [Background] Chittoodan S, Breen D, O'Donnell BD, Iohom G. Long versus short axis ultrasound guided approach for internal jugular vein cannulation: a prospective randomised controlled trial. Med Ultrason. 2011 Mar;13(1):21-5. PMID 21390339
- [Background] Phelan M, Hagerty D. The oblique view: an alternative approach for ultrasound-guided central line placement. J Emerg Med. 2009 Nov;37(4):403-8. doi: 10.1016/j.jemermed.2008.02.061. Epub 2008 Oct 1. PMID 18829208
- [Derived] Batllori M, Urra M, Uriarte E, Romero C, Pueyo J, Lopez-Olaondo L, Cambra K, Ibanez B. Randomized comparison of three transducer orientation approaches for ultrasound guided internal jugular venous cannulation. Br J Anaesth. 2016 Mar;116(3):370-6. doi: 10.1093/bja/aev399. Epub 2015 Dec 24. PMID 26705350
- See also: Web of the investigation project in navarrabiomed. Click here for more information about this study. — http://www.navarrabiomed.es

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The day before IJVC was to be performed, patients (aged 18 or above) in whom IJVC had been indicated were asked to participate in the study. Patients who did not meet any exclusion criteria were included.
Groups:
- Long Axis, In-plane Needle: Ultrasound-guided Internal jugular venous approach
  Long axis, in-plane needle:
  Jugular vein is ultrasonographically visualized in a longitudinal fashion (long axis) and the needle is inserted in the same ultrasound plane, aligned with the longitudinal axis of the transducer.
  Ultrasound-guided Internal jugular venous approach: The physician will use an ultrasound machine to perform an ultrasound-guided internal jugular venous cannulation: the needle and the vein will be visualized in real time in the ultrasound image to make the cannulation process easier and safer.
  In each one of three study arms, however, the ultrasound approach will be different depending on the axis on wich the vein is visualized (longitudinal, transversal or oblique) and the way the needle enters the ultrasound plane (in-plane or out of plane).
- Short Axis, Out-of-plane Needle: Ultrasound-guided Internal jugular venous approach
  Short axis, out-of-plane needle:
  Jugular vein is ultrasonographically visualized in a transverse fashion (short axis) and the needle is inserted perpendicular to the longitudinal axis of the transducer (out-of-plane).
  Ultrasound-guided Internal jugular venous approach: The physician will use an ultrasound machine to perform an ultrasound-guided internal jugular venous cannulation: the needle and the vein will be visualized in real time in the ultrasound image to make the cannulation process easier and safer.
  In each one of three study arms, however, the ultrasound approach will be different depending on the axis on wich the vein is visualized (longitudinal, transversal or oblique) and the way the needle enters the ultrasound plane (in-plane or out of plane).
- Oblique Axis, In-plane Needle: Ultrasound-guided Internal jugular venous approach
  Oblique axis, in-plane needle:
  Jugular vein is ultrasonographically visualized in an oblique axis (intermediate view between long and short axis) and the needle is inserted in the same ultrasound plane, aligned with the longitudinal axis of the transducer.
  Ultrasound-guided Internal jugular venous approach: The physician will use an ultrasound machine to perform an ultrasound-guided internal jugular venous cannulation: the needle and the vein will be visualized in real time in the ultrasound image to make the cannulation process easier and safer.
  In each one of three study arms, however, the ultrasound approach will be different depending on the axis on wich the vein is visualized (longitudinal, transversal or oblique) and the way the needle enters the ultrasound plane (in-plane or out of plane).
Period: Overall Study
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Started | 75 | 73 | 72
Completed | 75 | 73 | 72
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle | Total
Number analyzed (Participants) | 75 | 73 | 72 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13.6) | 64.9 (13.6) | 65.2 (15.0) | 64.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 29 | 83
  Male | 49 | 45 | 43 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 75 | 73 | 72 | 220
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 75 | 73 | 72 | 220
Cannulated IJV diameter (cm) [Mean (Standard Deviation); unit: centimeters (cm)] | 1.23 (0.3) | 1.20 (0.3) | 1.10 (0.2) | 1.20 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Cannulation Success
Description: Cannulation will be considered as "successful" once a flexible guidewire has been inserted into the internal jugular vein during the first 180 seconds from the moment the Seldinger needle pierces the skin. If time spent until guidewire insertion is more than 180 seconds, or if guidewire cannot be inserted into the internal jugular vein chosen, cannulation will be considered "unsuccessful". This outcome measure will be registered at the end of the cannulation process.
Time Frame: At the end of the cannulation process (180 seconds, maximum)
Measure: Number; unit: participants
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Number analyzed (Participants) | 75 | 73 | 72
participants | 73 | 71 | 68

2. Secondary Outcome: Number of Cannulation Attempts
Description: Number of cannulation attempts that have taken place before cannulation success. Any withdrawal of the needle followed by an advance will be considered a separated cannulation attempt.This outcome measure will be registered at the end of the cannulation process.
Time Frame: At the end of the cannulation process (180 seconds, maximum)
Measure: Mean (Standard Deviation); unit: attempts
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Number analyzed (Participants) | 75 | 73 | 72
attempts | 1.92 (1.36) | 1.51 (0.97) | 1.37 (0.84)

3. Secondary Outcome: First Attempt Cannulation
Description: Any cannulation that has been accomplished with a single cannulation attempt will be considered a "first attempt cannulation". This outcome measure will be registered at the end of the cannulation process.
Time Frame: At the end of the cannulation process (180 seconds, maximum)
Measure: Number; unit: participants
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Number analyzed (Participants) | 75 | 73 | 72
participants | 39 | 51 | 53

4. Secondary Outcome: Cannulation Time
Description: Time elapsed (seconds) from the moment the Seldinger needle pierces the skin to the moment the guidewire is inserted inside the vein. This outcome measure will be registered at the end of the cannulation process.
Time Frame: At the end of the cannulation process (180 seconds, maximum)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Number analyzed (Participants) | 75 | 73 | 72
seconds | 46.1 (36.3) | 35.0 (23.4) | 41.2 (23.9)

5. Secondary Outcome: Mechanical Complications
Description: The incidence of the following mechanical complications will be registered: number of patients with accidental arterial puncture, number of patients with puncture site bleeding, number of patients with puncture site haematoma, number of patients with pneumothorax, number of patients catheter tip misplacement. This outcome measure will be registered at the end of the cannulation process, and once a control chest x-Ray has been performed.
Time Frame: At the end of the cannulation process (180 seconds, maximum)
Measure: Number; unit: participants
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Number analyzed (Participants) | 75 | 73 | 72
participants | 3 | 11 | 5

6. Secondary Outcome: Infectious Complications
Description: The incidence of bacterial catheter colonization and catheter-related blood stream infection will be registered once the central venous catheter has been withdrawn. Patients will be followed for the duration of central venous access, an expected average of 8 weeks. The number of patients with bacterial colonization and catheter-related blood stream infection will be registered.
Time Frame: Once the central venous catheter is withdrawn (2 months)
Measure: Number; unit: participants
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Number analyzed (Participants) | 75 | 73 | 72
participants | 2 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Long Axis, In-plane Needle | Short Axis, Out-of-plane Needle | Oblique Axis, In-plane Needle
Serious Adverse Events (participants affected / at risk) | 2/75 | 0/73 | 0/72
Other Adverse Events (participants affected / at risk) | 5/75 | 11/73 | 5/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Long Axis, In-plane Needle (N=75) | Short Axis, Out-of-plane Needle (N=73) | Oblique Axis, In-plane Needle (N=72)
Catheter-related blood stream infection (Infections and infestations) | 2 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Long Axis, In-plane Needle (N=75) | Short Axis, Out-of-plane Needle (N=73) | Oblique Axis, In-plane Needle (N=72)
Posterior internal jugular venous wall puncture (Vascular disorders) | 0 | 8 | 1
Puncture site bleeding (Blood and lymphatic system disorders) | 1 | 2 | 0
Local cervical haematoma (Blood and lymphatic system disorders) | 2 | 1 | 2
Catheter misplacement (Vascular disorders) | 2 | 0 | 2

LIMITATIONS AND CAVEATS:
Results may be only extrapolative to experienced cannulators

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No